CLINICAL TRIAL: NCT02639078
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Single Ascending Dose Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TD-0714 in Healthy Subjects
Brief Title: Single Ascending Dose Study of TD-0714 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0139
Record Dates: First submitted 2015-11-25; First posted 2015-12-24 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Single ascending dose; volunteers; Phase 1; first-in-human; TD-0714

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TD-0714 (Experimental): One time dosing in capsule formulation
  Interventions: Drug: TD-0714
- Placebo (Placebo Comparator): Placebo comparator one time dosing in capsule formulation
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: TD-0714 — One time dosing in capsule formulation
  Arms: TD-0714
Drug: Placebo Comparator — One time dosing in capsule formulation
  Arms: Placebo

SUMMARY:
Single ascending dose study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of TD-0714 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 18 to 32 kg/m2 inclusive
* Women of child bearing potential must have a negative pregnancy test and either abstain from sex or use highly effective methods of birth control
* Women of non-childbearing potential are at least 2 years postmenopausal or are surgically sterile
* Males must abstain from sex or use highly effective methods of birth control
* Negative for HIV, and Hepatitis A, B, and C

Exclusion Criteria:

* Female subjects who are pregnant, lactating, breastfeeding or planning to become pregnant during the study.
* Subjects with a history of angioedema.
* Subject has evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
* Subject has acute illness (gastrointestinal, infection [e.g., influenza] or known inflammatory process)
* Subject bradycardia
* Subject has hypertension
* Subjects has orthostatic hypotension
* Subjects has orthostatic tachycardia
* Subject has a known personal or family history of congenital long QT syndrome or known family history of sudden death.
* Subject has donated blood or blood components or has had blood loss exceeding 400 mL within the 90 days prior to Screening.
* Additional exclusion criteria apply

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TD-0714 by assessing the number, severity and type of adverse events, including changes in vital signs, physical and neurological examinations, laboratory safety tests and ECGs | From Day 1 through end of study (Day 10)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of TD-0714 in plasma after a single-dose (SD): peak plasma concentration (Cmax) | Day 1 through end of study (Day 10)
PK of TD-0714 in plasma after a SD: time to peak plasma concentration (Tmax) | Day 1 through end of study (Day 10)
PK of TD-0714 in plasma after a SD: time to last measurable concentration (Tlast) | Day 1 through end of study (Day 10)
PK of TD-0714 in plasma after a SD: area under the plasma concentration vs. time curve from time zero to the last quantifiable concentration (AUC0-t) | Day 1 through end of study (Day 10)
PK of TD-0714 in plasma after a SD: area under the plasma concentration vs. time curve from time zero to 24 hours postdose (AUC0-24) | The day before dosing (Day -1) to the day after dosing (Day 2)
PK of TD-0714 in plasma after a SD: area under the plasma concentration vs. time curve from time zero to infinity (AUC0-∞) | Day 1 through end of study (Day 10)
PK of TD-0714 in plasma after a SD: CL/F (oral plasma clearance) | Day 1 through end of study (Day 10)
PK of TD-0714 in plasma after a SD: Vz/F (apparent volume of distribution during the terminal phase) | Day 1 through end of study (Day 10)
PK of TD-0714 in plasma after a SD: t1/2 (half-life) | Day 1 through end of study (Day 10)
PK of TD-0714 in urine after a SD: Ae (amount excreted in urine) | Day 1 through end of study (Day 10)
PK of TD-0714 in urine after a SD: Fe (fraction of oral dose excreted in urine) | Day 1 through end of study (Day 10)
PK of TD-0714 in urine after a SD: Clr (renal clearance) | Day 1 through end of study (Day 10)

OTHER OUTCOMES:
Pharmacodynamics assessments for plasma atrial natriuretic peptide (ANP) concentrations | The day before dosing (Day -1) to the day after dosing (Day 2)
Pharmacodynamics assessments for urine atrial natriuretic peptide (ANP) concentrations | The day before dosing (Day -1) to the day after dosing (Day 2)
Pharmacodynamics assessments for plasma cyclic guanosine monophosphate (cGMP) concentrations | The day before dosing (Day -1) to the day after dosing (Day 2)
Pharmacodynamics assessments for urine cyclic guanosine monophosphate (cGMP) concentrations | The day before dosing (Day -1) to the day after dosing (Day 2)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Celerion, Lincoln, Nebraska, United States